CLINICAL TRIAL: NCT04496037
Title: Mechanistic Evaluation of Treatments for Acute Antibody-Mediated Rejection of the Kidney Transplant
Acronym: MOT-AMR
Status: Not yet recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: University of Cambridge (Other); Viapath LLP (Unknown)
Responsible Party: Sponsor
Other Study IDs: 19HH5204
Record Dates: First submitted 2020-07-29; First posted 2020-08-03 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Transplant; Complication, Rejection
MeSH Terms: conditions — Rejection, Psychology | interventions — Rituximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Enrolment and indication renal transplant biopsies: material left over after diagnosis Optional renal transplant protocol biopsy Leftover serum from samples taken at time of biopsy Extra blood sample taken at time of biopsy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard of care (SOC): See NCT03994783
- Rituximab + SOC (SOCR): See NCT03994783
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — See NCT03994783
  Groups: Rituximab + SOC (SOCR)

SUMMARY:
The best treatment for kidney failure is a kidney transplant, but a transplanted kidney only works for about 10 to 15 years on average. One of the reasons that a transplanted kidney can stop working is that the body develops antibodies against it. Antibodies are proteins produced by the body to fight infections. They play a vital role in dealing with infection but in some transplant patients they can 'fight' the organ, meaning it could stop working. This is called acute antibody-mediated rejection (AAMR). A patient experiencing AAMR can be treated to extend the life of the transplanted kidney, but the chances of the kidney still working 4 years later are reduced. There is currently a clinical trial for UK kidney transplant patients who develop AAMR, called TAR:GET-1. Patients participating in TAR:GET-1 will either receive the standard treatment that is currently given in this situation, or the standard treatment with the addition of rituximab. TAR:GET-1 will answer the question: does adding rituximab to standard treatment lengthen the life of a kidney transplant? A second, sub-study is being proposed of the patients enrolled in TAR:GET-1, that will use the existing blood and biopsy samples already taken during TAR:GET-1 plus an optional extra biopsy of the kidney transplant, to improve our understanding of how the treatments of AAMR work. Patients enrolled in TAR:GET-1 will have had a blood test and biopsy of the transplanted kidney to establish the diagnosis of AAMR. They will also have had further blood tests after treatment, and may also have further biopsies taken if their clinician needs these as part of normal care. Material left over in these samples can be used to analyse how treatment works. In addition, patients will be asked if they agree to an extra biopsy of the transplanted kidney 6 months after the treatment begins. These samples will be analysed at a deeper level than would normally be done, looking at the antibodies and biopsies in detail to answer 2 key questions: 1) Can the unique characteristics noted in an individual patient's antibodies and biopsy predict whether a kidney transplant will be lost as a result of AAMR?; 2) Can we tell treatment is working by looking at the changes in a patient's antibodies and biopsies before and after treatment? The answers to these questions will help us understand AAMR and how its treatments work, and potentially improve our ability to select the right treatment for the right patients.

DETAILED DESCRIPTION:
Design: Prospective observational study of patients enrolled in TAR:GET-1

Objectives: TAR-GET-1 (starting in 2019) is a multi-centre UK clinical trial that will compare standard of care (SOC) treatment of Acute Antibody-Mediated Rejection of the Kidney Transplant (AAMR) to standard of care plus rituximab (SOCR). This trial presents a rare opportunity to investigate the mechanisms of action of treatments (including rituximab) in AAMR. The rationale for using rituximab is the depletion of CD20-positive precursors to antibody-producing cells. However, rituximab has effects on other B cell subtypes and not all studies have shown antibody level reductions. Furthermore, AAMR is a heterogeneous disease, as defined by variability in mechanistic markers of AAMR in blood (B cell and antibody characteristics) and in transplant biopsies (histological features and gene expression).

The objectives of this study are:

1. To investigate how treatment with rituximab affects these mechanistic markers, by comparing SOC to SOCR
2. To predict treatment benefit early, by analysing the effect of treatment on the mechanistic markers

Methodology: In patients enrolled in TAR:GET-1 (n=170), mechanistic markers will be analysed with established proof of concept (B cell and antibody characteristics, histological and transcriptional markers in the biopsy) at baseline and on follow-up, making use of clinical data, surplus diagnostic material from TAR:GET-1, and material from optional extra blood samples for research taken as part of TAR:GET-1, at 3,6 and 12 months. An optional protocol biopsy at 6 months post treatment will also be offered.

TARGET-1 is assessing DSA MFI and target and B lymphocyte numbers at baseline and 3 months post-treatment. This study will in addition analyse:

1. Serum DSA MFI and target at 6 months; complement-activating ability at baseline, 3 months and 6 months;
2. Biopsy Banff histological scores at baseline and in post-treatment indication biopsies and an optional protocol biopsy;
3. Biopsy AAMR-related transcript signature, assessed using Nanostring nCounter technology, at baseline and in post-treatment biopsies indication biopsies and an optional protocol biopsy;
4. B lymphocyte numbers at 6 months.

Differences pre- and post-treatment will be analysed comparing SOC and SOCR. Mediation analysis models will be used to decompose total effect of treatment effect on graft loss at 4 years (primary end point) into an indirect effect, which measures how much of the effect acts through the intermediate variable(s), and a residual direct effect.

Number of Subjects and Study populations: 170 subjects enrolled in TAR:GET-1

Outcome measures: same as primary outcome of TAR:GET-1 (graft loss at 4 years after initiation of treatment)

Inclusion Criteria: All patients enrolled in TAR:GET-1 ; Signed informed consent prior to any study specific procedures.

Exclusion Criteria: None

Duration of study: 8 years (duration is dictated by the need for primary outcome of TAR-GET-1 to be reached)

Statistical Methods: Data from this research project will be merged and linked with data from the TAR:GET-1 clinical trial by the statistician team.

Descriptive data: This will include description of all the biological characteristics analysed in 2 populations (rituximab + SOC and SOC) at baseline and at all follow-up time points. Summary statistics (mean, median, SD, range for continuous variables, and frequency tables for categorical variables) will be reported broken down by treatment, with exploratory figures (box-and-whisker plots for continuous, and stacked bar-charts for categorical).

Outcome analysis: Appropriate measures of differences between treatment groups will be estimated with point estimates, 95% confidence intervals, and p-values. Depending on the type of variable (continuous, categorical, time-to-event), regression techniques (linear, logistic, cox) and transformation of the endpoints will be considered.

Differences in characteristics comparing pre- to post-treatment samples at sequential time points will be analysed comparing the 2 groups of patients (SOCR versus SOC) using r mixed effect models repeat measurement techniques.

Mediation analysis, a special case of regression analysis, will be used to document that the treatment effects a change in the biomarker. Mediation analysis models will be used to decompose total effect of treatment effect on graft loss into an indirect effect, which measures how much of the effect acts through the intermediate variable(s), and a residual direct effect. All the mediation analyses will be based on the Intention-to-Treat principle. The same form of outcome models will be fitted as for the efficacy analyses, including the mediator as a covariate. The mediation package within R will be used which was developed specifically to make valid causal inference in explanatory analyses of the mechanisms of treatment-induced change in clinical outcomes in randomised clinical trials. All estimates of treatment differences will be summarised using effect size estimates and 95% confidence intervals (Dunn 2013). Collaborator for mediation analysis: Prof Ian White, Professor of Statistical Methods for Medicine, UCL.

ELIGIBILITY:
Inclusion Criteria:

All patients enrolled in TAR:GET-1 Signed informed consent prior to any study specific procedures.

Exclusion Criteria:

None

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients enrolled in TAR:GET-1
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Allograft Survival as assessed by statistical model | 4 years
  Statistical model measuring allograft survival as defined as duration from the date of randomisation to the date of eGFR ≤15 mL/min/1.72 m2, or the date of renal replacement therapy (date of starting dialysis dependency, transplantation etc), whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Candice Roufosse, MD PhD, Principal Investigator — Imperial College London

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2020-05-27): https://cdn.clinicaltrials.gov/large-docs/37/NCT04496037/Prot_000.pdf